CLINICAL TRIAL: NCT04220710
Title: Methylation of cfDNA in Diagnosis and Differential Diagnosis of Ovarian Endometriosis
Brief Title: cfDNA in Diagnosis and Differential Diagnosis of Ovarian Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, shuwang, Associate Professor, Peking Union Medical College Hospital
Other Study IDs: MCFD
Record Dates: First submitted 2020-01-04; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Circulating Free DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and FFPF samples in marker selection group; blood samples in marker validation group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Marker selection group: Methalation detection of circulating free DNA and FFPF samples from pathologically confirmed patients with ovarian endometriosis(30 cases), ovarian cancer (30 cases)and other benign ovarian tumors (30 cases)will be performed to select markers for ovarian endometriosis diagnosis.
  Interventions: Diagnostic Test: DNA extraction and methylation detection
- Marker validation group: The selected markers will be validated in patients with ovarian cysts (300 cases )found by ultrasound. The diagnosis accuracy of the markers will be evaluated by comparing with the pathological diagnosis.
  Interventions: Diagnostic Test: DNA extraction and methylation detection

INTERVENTIONS:
Diagnostic Test: DNA extraction and methylation detection — DNA extraction and methylation detection

SUMMARY:
Methylation detection of circulating free DNA to identify markers for diagnosis and differential diagnosis of ovarian endometriosis.

DETAILED DESCRIPTION:
Methylation detection of circulating free DNA and FFPF samples from patients with ovarian endometriosis, ovarian cancer and other benign ovarian cysts will be performed to select markers for ovarian endometriosis diagnosis. The markers will be validated in patients with ovarian cysts found by ultrasound. The diagnosis accuracy of the markers will be evaluated by comparing with the pathological diagnosis.

ELIGIBILITY:
1. Marker selection group:

1. patients with ovarian endometriosis:

   Inclusion Criteria:
   1. pathologically diagnosed as ovarian endometriosis;
   2. surgery was performed in PUMCH

      Exclusion Criteria:

   a. combined with other gynecological benign and malignant tumors; b. clinically suspected malignant tumors; c. combined with other systemic malignancies or malignancies history; d. pregnant patients
2. patients with ovarian cancer:

Inclusion Criteria:

1. pathologically diagnosed as epithelial ovarian cancer;
2. surgery was performed in PUMCH

Exclusion Criteria:

1. combined with gynecological benign tumors and other malignant tumors;
2. combined with other systemic malignancies or malignancies history;
3. pregnant patients (3) patients with other benign ovarian tumors:

Inclusion Criteria:

1. pathologically diagnosed as benign ovarian tumors but not ovarian endometriosis;
2. surgery was performed in PUMCH

Exclusion Criteria:

a. combined with other gynecological benign and malignant tumors; b. clinically suspected malignant tumors; c. combined with other systemic malignancies or malignancies history; d. pregnant patients

2. Marker validation group:

Inclusion Criteria:

1. ovarian cysts found through ultrasound ;
2. surgery will be performed in PUMCH

Exclusion Criteria:

1. combined with other gynecological benign and malignant tumors;
2. clinically suspected malignant tumors;
3. combined with other systemic malignancies or malignancies history;
4. pregnant patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Marker selection group: patients with ovarian endometriosis, ovarian cancer and other benign ovarian tumors
  2. Marker validation group: patients with ovarian cysts found through ultrasound ;
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-02-20 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
The efficacy of cfDNA methylation in the diagnosis of ovarian endometriosis | 12 months
  The sensitivity, specificity and accuracy are calculated according to standard definitions to evaluate the efficacy of cfDNA methylation in the diagnosis of ovarian endometriosis

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China